CLINICAL TRIAL: NCT03487614
Title: Evaluation of a Primary Care Weight Management Program in Children Aged 2 to 5 Years: Changes in Feeding Practices, Health Behaviors, and Adiposity
Brief Title: Evaluation of a Primary Care Weight Management Program in Children Aged 2 to 5 Years
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Corewell Health West (Other)
Collaborators: Blue Care Network of Michigan (Other); We Are For Children, LLC (Unknown)
Responsible Party: Principal Investigator, Jared Tucker, Epidemiologist, Corewell Health West
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WAFC25
Record Dates: First submitted 2018-03-21; First posted 2018-04-04 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Childhood Obesity; Feeding Behavior; Physical Activity
Keywords: pediatric obesity; preschool children; non-responsive feeding; body mass index; parenting
MeSH Terms: conditions — Pediatric Obesity; Feeding Behavior; Motor Activity

STUDY DESIGN:
Intervention Model Description: We Are for Children, LLC (WAFC), is a collaboration of non-profit pediatric practices in West Michigan formed to help members respond to healthcare needs. Four primary care pediatric offices from WAFC were selected to participate in the current study based on site interest and capacity. Participating pediatric offices were then matched into pairs based on similarities in office size (i.e. physician FTEs and patient load) and patient demographics characteristics, after which one of each matched pair was assigned as a treatment or control site.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavior-based parental intervention (Experimental): The study intervention included two primary components: 1) physician-family health behavior conversations during well-child visits, and 2) four monthly visits with a RDN to evaluate, educate, and implement improved feeding habits and nutritional choices. A third optional component of the intervention included counseling sessions with a social worker to help families overcome barriers to change, such as food security, family relationships, and general parenting strategies.
  Interventions: Behavioral: Behavior-based parental intervention
- Control (No Intervention): Control parents signed the informed consent document and then completed all baseline assessments during their child's medical visit. Control participants then received their usual medical care. Follow-up evaluations, including child anthropometry and completion of study surveys were assessed approximately 6 months later during a second office visit. For children <3 years of age at baseline, follow up visits coincided with their subsequent well-child visit (i.e. 30-month or 3-year appointment) as per AAP visit frequency recommendations. For patients ≥3 years of age, families attended a separate office visit 6 months after their baseline visit in order to complete follow-up study assessments.

INTERVENTIONS:
Behavioral: Behavior-based parental intervention — Behavioral intervention designed to promote healthy feeding behaviors in parents of 2-5 year olds, and to modify parenting practices in a way that encourages adequate physical activity, sufficient sleep, and healthy nutrition, while limiting sedentary behaviors.
  Arms: Behavior-based parental intervention

SUMMARY:
Primary care offers a promising setting for promoting parenting practices that shape healthy eating and physical activity behaviors of young children. This study assessed the impact of a parent-based, primary care intervention on the feeding habits, health behaviors, and body mass index (BMI) of 2-5 year olds with elevated or rapidly-increasing BMI. Four private pediatric offices in West Michigan were assigned as control (n=2) or intervention (n=2) sites based on patient load and demographics. Treatment families were recruited at well-child visits to receive physician health-behavior counseling and four visits with a registered dietitian nutritionist (RDN) over a 6-month period. Outcomes included percent of the 95th BMI percentile (%BMI95), the Family Nutrition and Physical Activity survey (FNPA), and the Feeding Practices and Structure Questionnaire (FPSQ).

ELIGIBILITY:
Inclusion Criteria:

* Age between 2 and 5 years
* BMI ≥85th percentile for age and sex, using the 2000 CDC growth chart, or BMI percentile increase within the past year equivalent to crossing at least two growth chart lines per year on a standard CDC growth chart, excluding the 5th percentile (e.g., 10th & 25th, 25th & 50th, 50th & 75th, 75th & 85th). This rate of increase is equivalent to ≥0.67 standard deviations per year (BMI z-score), and, when occurring in this age group, has been shown to increase risk of adult obesity

Exclusion Criteria:

* Known disorder of the HPA axis
* Use of glucocorticoid medication
* Non-English speaking

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 184 (Actual)
Dates: Start 2014-07-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Anthropometry | Change from baseline to follow-up at 6 months
  Age- and sex-specific body mass index such as percent of the 95th BMI percentile
FNPA | Change from baseline to follow-up at 6 months
  Family Nutrition and Physical Activity screening tool
FPSQ | Change from baseline to follow-up at 6 months
  Feeding Practices and Structure Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Jared M Tucker, PhD, Principal Investigator — Corewell Health West

IPD SHARING:
Plan to Share IPD: No
Data sharing is a possibility upon approval from IRB.